CLINICAL TRIAL: NCT00908180
Title: A Phase II Study of Reduced Intensity Allogeneic Transplantation for Refractory Hodgkin Lymphoma
Brief Title: Carmustine, Etoposide, Cytarabine, Melphalan, and Alemtuzumab Followed by Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CRUK-PAIReD; CDR0000640493 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2008-004956-60; EU-20930; UCL/08/0121
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Alemtuzumab; Carmustine; Cyclosporine; Cytarabine; Etoposide; Melphalan

INTERVENTIONS:
Biological: alemtuzumab
Biological: donor lymphocytes
Drug: carmustine
Drug: cyclosporine
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. Monoclonal antibodies, such as alemtuzumab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine before and after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

PURPOSE: This phase II trial is studying the side effects of giving carmustine together with etoposide, cytarabine, melphalan, and alemtuzumab followed by donor stem cell transplant and to see how well it works in treating patients with relapsed or refractory Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To document the toxicity and feasibility of reduced-intensity conditioning regimen comprising carmustine, etoposide, cytarabine, melphalan, and alemtuzumab followed by allogeneic hematopoietic stem cell transplantation in patients with primary refractory or relapsed Hodgkin lymphoma.
* To document the survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Conditioning regimen: Patients receive BEAM chemotherapy comprising carmustine IV over 2 hours on day -6, etoposide IV over ≥ 1 hour on days -5 to -2, cytarabine IV over 15 minutes twice daily on days -5 to -2, and melphalan IV on day -1. Patients also receive alemtuzumab IV on days -5 to -1.
* Allogeneic hematopoietic stem cell transplantation (HSCT): Patients undergo allogeneic HSCT on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV (or orally once tolerable) beginning on day -1 and continuing until day 60, followed by a taper in the absence of GVHD.
* Donor lymphocyte infusion (DLI): Patients with mixed chimerism or stable residual disease at 6 months after HSCT or disease progression or relapse at any time after HSCT may receive DLI in the absence of GVHD.

After completion of study treatment, patients are followed periodically for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of Hodgkin lymphoma, meeting 1 of the following criteria:

  * Refractory to initial multi-agent induction therapy and achieved less than a complete response to one line of salvage chemotherapy
  * In first relapse and achieved less than a partial response to one line of salvage chemotherapy
* No progressive disease
* Must have an HLA-matched (≥ 9/10) sibling or unrelated donor available

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Creatinine clearance ≥ 50 mL/min
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* LVEF ≥ 40%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2-3 months after completion of study treatment
* No HIV positivity
* No other malignancy within the past 5 years, except for nonmelanoma skin cancer or stage 0 (in situ) cervical carcinoma
* No concurrent serious medical condition that would preclude an allograft
* No symptomatic respiratory compromise

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior high-dose therapy or allograft

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 3 years

SECONDARY OUTCOMES:
Donor engraftment rates, including chimerism at 3 and 6 months
Non-relapse mortality at 100 days, 1 year, and 2 years post-transplant
Incidence of grade II-IV toxicity as assessed by NCI CTCAE v3.0
Incidence, severity, and timing of acute and chronic graft-versus-host disease
Response rates
Relapse rates
Response to donor lymphocyte infusions
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peggs, MD, Principal Investigator — University College London (UCL) Cancer Institute

REFERENCES:
- [Derived] Das-Gupta E, Thomson KJ, Bloor AJC, Clark AD, Mackinnon S, Kayani I, Clifton-Hadley L, Patrick P, El-Mehidi N, Lawrie A, Kirkwood AA, Russell NH, Linch DC, Peggs KS. Allo-HSCT in transplant-naive patients with Hodgkin lymphoma: a single-arm, multicenter study. Blood Adv. 2019 Dec 23;3(24):4264-4270. doi: 10.1182/bloodadvances.2019001016. PMID 31869413